CLINICAL TRIAL: NCT02406326
Title: A Prospective Evaluation of BioMime™ - Sirolimus Eluting Coronary Stent in a Multi- Centre Study.
Brief Title: An Evaluation of BioMime™ - Sirolimus Eluting Coronary Stent in a Multi- Centre Study.
Acronym: meriT-2
Status: Completed | Type: Observational
Sponsor: Meril Life Sciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: BIO1TR/MLS/100209
Record Dates: First submitted 2015-03-30; First posted 2015-04-02 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a multi centre, prospective trial. 250 patients will be enrolled in the study.(10 patients per centre involving approximately 25 centres). Patients will be followed up clinically for twelve months post-procedure at 1 month, 6 months & 12 months. All patients will have a repeat angiography at 8 months. Clinical follow-up will be maintained for years 3 & 5 post-implant.

DETAILED DESCRIPTION:
This is a multi centre, prospective observational study. 250 patients will be enrolled in the study. 10 patients per centre involving approximately 25 centres. All the patients will be followed for twelve months post-procedure. All patients will have a repeat angiography assessment at 8 months. An additional clinical follow-up will be maintained for years 3 & 5 post-implant.

Approximately 250 patients with obstructive coronary artery disease with a vessel size between ≥2.5 to ≤3.5 mm in diameter by visual estimate and who meet all eligibility criteria will be treated with the Sirolimus Eluting Stent.

It is anticipated that the total length of the study will be 16 months: 4 months to complete patient enrollment and 12 months for angiographic follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be ≥18 years of age;
2. Patient is an acceptable candidate for PTCA, Stenting, or Emergent CABG;
3. Symptomatic ischemic heart disease (CCS class 1-4 , Braunwald class IB, IC, IIB, IIC,IIIB,IIIC) and/or objective evidence of myocardial ischemia;
4. TIMI (Thrombolysis In Myocardial Infarction) flow grade ≥ 2 ;
5. C.T.O's (Chronic Total Occlusions) and Bifurcation Lesions may also be attempted;
6. Target lesion stenosis is >50% and <100% ;
7. Target lesions are de novo;
8. Target lesions ≤ 35mm in length (by visual estimation) that can be treated (covered) by one single study stent (13 to 40mm in length)
9. Target lesion located in a major epicardial coronary vessel with reference of ≥ 2.5 - ≤ 3.5mm in diameter (by visual estimation)
10. Target lesions which can be covered by one stent, no overlapping allowed (lesion stent ratio of at least 1.5)
11. The patient and/or his legal representative has been informed of the nature of the study and agrees to its provisions and has provided a written informed consent.

Exclusion Criteria:

General exclusion criteria:

1. Women of childbearing potential;
2. Impaired renal function (creatinine > 2.0 mg/dl or 180 μmol/l);
3. Any patient who has a platelet count < 100,000 cells/mm3 or > 700,000 cells/mm3, a WBC of < 3,000 cells/mm3, or documented or suspected liver disease (including laboratory evidence of Hepatitis;
4. Recipient of an organ (Heart, Kidney, Lung or Liver) transplant;
5. History of CVA or TIA within the last 3 months
6. Patient with a concomitant disease having a life expectancy of less than 12 months;
7. Known allergies or contraindication to mTOR inhibitor class of drugs (Sirolimus), Aspirin, Clopidogrel Bisulphate (Plavix®), Heparin, Cobalt Chromium/Nickel, contrast media;
8. Any significant medical condition which in the investigator's opinion may interfere with the patient's optimal participation in the study such as an active infection or peptic ulcer or upper GI bleeding;
9. Currently participating in an investigational drug or another device study, or subject to inclusion in another investigational drug or another device study during follow-up.
10. Clinically relevant contraindication to aspirin, heparin, clopidogrel bisulphate, including thrombocytopenia, neutropenia, or leukopenia
11. Patients with Cardiogenic Shock.

Angiographic Exclusion criteria:

1. Left main coronary artery disease with ≥ 50% stenosis,
2. Angiographic evidence of thrombus (thrombus larger than half the diameter of the vessel and/or requiring other adjunctive interventions such as Angiojet, Exciser, Thrombolysis, etc.),
3. Left Ventricular Ejection Fraction ≤30 %,
4. Saphenous Vein Graft Interventions, (S.V.G's)
5. Patients presenting with an ongoing Acute Myocardial Infarction (AMI),
6. Patients having undergone a PCI within 48 hours of an AMI episode.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of 250 patients with an obstructive coronary artery disease with few exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2009-08-27 (Actual); Primary Completion 2016-12-27 (Actual); Study Completion 2016-12-27 (Actual)

PRIMARY OUTCOMES:
Major Adverse Cardiac Events (MACE) days | 30 days
  composite of Death, MI (both Q-wave and Non Q-wave MI), Emergent CABG, or Clinically driven TLR (repeat PCI or CABG) and measured percentage wise

SECONDARY OUTCOMES:
Major Adverse Cardiac Events (MACE) | Until 12 months
  Major adverse cardiac events is defined as the aggregate of cardiac death, myocardial infarction (MI) attributed to target vessel, and any target lesion revascularization (TLR)
Device related SAEs | Until 12 months
  Serious Adverse Events
Angioghraphic stent thrombosis | After 30 days until 12 months
  Acute (In hospital), Subacute (post procedure until 30 days) and Late (after 30 days until 12 months)
Angiographic/Device success, Procedural Success, Clinically justified Target Lesion Revascularization | At 12 months
  Quantitative Coronary Angiography derived vessel parameters In stent and 5 mm proximal and 5 mm distal from the edge of the stent (In-segment), Acute Gain (mm), Mild (%), Late loss (mm) and Binary Restenosis (%) rate, In stent MLD pre, post and 8 months angiographic follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Ashok Seth, FRCP, FACC,FMRCP, MBBS, Principal Investigator — Fortis Escorts Heart Institute & Research Centre; Dr. Ajit Mullasari, DNB, DM, MD, MBBS, Principal Investigator — Madras Medical Mission; Dr. Rohit M Kumar, DM, MD, MBBS, Principal Investigator — Advance Cardiac Centre; Dr. Samuel K Mathew, DM, MD, MBBS, Principal Investigator — Apollo Group of Hospitals; Dr. G S Wander, DM, MD, MBBS, Principal Investigator — Hero DMC Heart Institute; Dr. C. N. Manjunath, DM, MD, MBBS, Principal Investigator — Sri Jayadeva Institute of Cardiovascular Sciences & Research; Dr. Thomas Alexander, FCSI, FICC, FACC, DM, MD, MBBS, Principal Investigator — Kovai Medical Centre and Hospitals Ltd; Dr. Suresh Vijan, MRCP, MD, MBBS, Principal Investigator — Fortis/Wockhardt Hospital; Dr. Suhas Hardas, DM, MD, MBBS, Principal Investigator — Poona Hopsital & Research Centre; Dr. Sunitha Abraham, DNB, MD, MBBS, Principal Investigator — Narayana Hrudayalaya Institute of Medical Sciences; Dr. Prabhakar Shetty, FACC, DM, MD, MBBS, Principal Investigator — Columbia Asia Hospitals
Locations (11):
- India (11):
  - Columbia Asia Hospitals, Bangalore, Karnataka
  - Sri Jayadeva Institute of Cardiovascular Sciences & Research, Bangalore, Karnataka
  - Narayana Hrudayalaya Institute of Medical Sciences, Bangalore, Karnataka
  - Fortis/Wockhardt Hospital, Mumbai, Maharashtra
  - Poona Hopsital & Research Centre, Pune, Maharshtra
  - Fortis Escorts Heart Institute & Research Centre, New Delhi, National Capital Territory of Delhi
  - Advance Cardiac Centre, Chandigarh, Punjab
  - Hero DMC Heart Institute, Ludhiana, Punjab
  - Madras Medical Mission, Chennai, Tamil Nadu
  - Apollo Group of Hospitals, Chennai, Tamil Nadu
  - Kovai Medical Centre and Hospitals Ltd, Coimbatore, Tamil Nadu

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Study results at 12 month follow up — http://www.asiaintervention.org/asia-pacific-hotlines-at-tct-2015-bioresorbable-vascular-scaffolds-versus-metallic-stents-in-patients-with-coronary-artery-disease-absorb-china-trial/